CLINICAL TRIAL: NCT04895137
Title: Safety and Efficacy of mFOLFOX6+ Bevacizumab+PD-1 Monoclonal Antibody Treatment Combinations in Patients With Local Advanced Microsatellite Stability Colorectal Cancer --an Open Label, Multicenter, Prospective Phase Ⅱ Study (BASKETII)
Brief Title: mFOLFOX6+Bevacizumab+PD-1 Monoclonal Antibody in Local Advanced MSS CRC
Acronym: BASKETⅡ
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sixth Affiliated Hospital, Sun Yat-sen University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: E2021056
Record Dates: First submitted 2021-05-18; First posted 2021-05-20 (Actual); Last update posted 2025-01-22 (Actual); Status verified 2024-09

CONDITIONS: Colorectal Cancer; Immunotherapy
Keywords: Colorectal cancer; pMMR/MSS; PD-1 monoclonal antibody; Bevacizumab; mFOLFOX6
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- mFOLFOX6+ Bevacizumab+PD-1 monoclonal antibody treatment combinations (Experimental): mFOLFOX6+ Bevacizumab+PD-1 monoclonal antibody treatment combinations in patients with local advanced microsatellite stability colon and upper rectum cancer
  Interventions: Drug: mFOLFOX6+Bevacizumab+PD-1 monoclonal antibody treatment combinations

INTERVENTIONS:
Drug: mFOLFOX6+Bevacizumab+PD-1 monoclonal antibody treatment combinations — mFOLFOX6+ Bevacizumab+PD-1 monoclonal antibody treatment combinations in patients with local advanced microsatellite stability colorectal cancer
  Other Names: mFOLFOX6+Bevacizumab+Sintilimab treatment combinations

SUMMARY:
Immunotherapy has achieved significant therapeutic effect in DNA mismatch repair-deficient or microsatellite instability-high (dMMR/MSI-H) colorectal cancer (CRC). However, for proficient mismatch repair(pMMR)/microsatellite stable(MSS) CRC, the curative effect of PD-1 monoclonal antibody was poor and most of the data came from stage Ⅳ patients with distant metastasis. Among the whole CRC patients, more than eighty-five percent were pMMR/MSS CRC. It would be very inspiring when major CRC patients(pMMR/MSS) could be benefit from immunotherapy. For T4NxM0 CRC patients, R0 resection was difficult to achieve. If the patients could not got R0 resection, which means the tumors were almost destined to recurrent and patients life time were counting down. Whether combined treatment of mFOLFOX6+ Bevacizumab+PD-1 monoclonal antibody could maximize the curative effect was still unknown. This study aims to evaluate the effect and safety of mFOLFOX6+ Bevacizumab+PD-1 monoclonal antibody treatment combinations in patients with local advanced(T4NxM0) pMMR/MSS CRC.

DETAILED DESCRIPTION:
Immunotherapy has achieved significant therapeutic effect in DNA mismatch repair-deficient or microsatellite instability-high (dMMR/MSI-H) colorectal cancer (CRC). MMR expression and MSS status are the important effective factors of immunotherapy. PD-1monocolnal antibody therapy has accessed excellent treatment effect in advanced dMMR/MSI-H CRC and neoadjuvant therapeutic effect in early colon cancer, more than fifty percent of dMMR/MSI-H CRC patients might get pathological complete response(pCR) after PD-1 monoclonal antibody treatment. The treatments had been proved to be safe and the toxicities were controllable. However, for proficient mismatch repair(pMMR)/microsatellite stable(MSS) CRC, the curative effect of PD-1 monoclonal antibody was poor and most of the data came from stage Ⅳ patients with distant metastasis. Among the whole CRC patients, more than eighty-five percent were pMMR/MSS CRC. It would be very inspiring when major CRC patients(pMMR/MSS) could be benefit from immunotherapy. For T4NxM0 CRC patients, R0 resection was difficult to achieve. If the patients could not got R0 resection, which means the tumors were almost destined to recurrent and patients life time were counting down. However, there were no standard conversion of neoadjuvant treatment recommendations for T4NxM0 CRC. Although PD-1 monoclonal antibody alone has poor effect in pMMR/MSS CRC, it seems to be effective in early stage of MSS CRC(Nicole study) or when it was combined with chemotherapy or target therapy. So far, whether combined treatment of mFOLFOX6+ Bevacizumab+PD-1 monoclonal antibody could maximize the curative effect was still unknown. This study aims to evaluate the effect and safety of mFOLFOX6+ Bevacizumab+PD-1 monoclonal antibody treatment combinations in patients with local advanced(T4NxM0) pMMR/MSS CRC.

ELIGIBILITY:
Inclusion Criteria:

* Histological identified colon and upper rectum adenocarcinoma, Tumor biopsy immunohistochemical (IHC) identified pMMR, including all of the MSH1,MSH2,MSH6 and PMS2 protein expression and diagnosed as proficient mismatch repair(pMMR), or next generation sequencing identified (MSS)； MRI identified tumor inferior margin higher than peritoneal reflection,
* Clinical staging T4NxM0, with or without positive MRF, with or without positive EMVI,
* Staging method：all patients undergo chest,abdominal and pelvic enhanced CT, rectal palpation, high resolution MRI examination，positive perienteric lymph node(LN): short diameter ≥10mm LN or LN with typical metastatic shape and MRI character, clinical data should be re-evaluated and judged by center evaluation group when there are contradictory stagings，distant metastasis were excluded by chest and abdominal enhanced CT and pelvic enhanced MRI,
* No intestinal obstruction symptom，or obstruction relieved after proximal colostomy,
* No rectal surgery history,
* No chemotherapy or radiotherapy history,
* No biopharmaceutical treatment history(such as monoclonal antibody), immunotherapy(such as anti PD-1antibody, anti PD-L1 antibody, anti PD-L2 antibody or anti CTLA-4), or other research drug treatment,
* Endocrinotherapy history restriction:No
* informed consent assigned,

Exclusion Criteria:

* Arrhythmia need anti-arrhythmia treatment(except β-blocking agent or Digoxin)，symptomatic coronary heart disease or myocardial ischemia(myocardial infarction within 6 months) or congestive heart-failure (CHF) > NYHA grade II,
* Severe hypertension not well controlled by drugs,
* HIV infection history or active phase of chronic Hepatitis B or C(high copies of virus DNA),
* Active tuberculosis(TB)，accepting anti-TB treatment or anti-TB treatment within 1 year before trial screen,
* Other active clinical severe infection(NCI-CTC V5.0),
* Outside pelvic distant metastasis evidences,
* Dyscrasia, organ dysfunction,
* Pelvic or abdominal radiotherapy history,
* Multiple CRC or Multi-primary tumors；
* Epilepsy need treatments(Steroid or anti-epilepsy therapy),
* Other malignant tumor history within 5 years,
* Over abuse of drugs, medical and psychological or social conditions that might interfere patients or evaluation of the study results,
* Any active autoimmune disease or autoimmune disease history (including but not restricted：interstitial pneumonia, uveitis,enteritis, hepatitis,hypophysitis, nephritis, hyperthyroidism, hypothyroidism, asthma need bronchodilators),
* Any anti-infection vaccine injection 4 weeks before inclusion ,
* Long-term exposure to immune-suppressor, combination of systemic or topical use of corticosteroids (dose>10mg/day prednisolone or equivalent hormone)；
* Known or suspicious allergy to any study related drugs,
* Any unstable state might cause damage to the safety and compliance of patients,
* Pregnant or breast feeding women who has ability to have children while without contraception,
* Refuse to sign informed consent

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2021-05-01 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2024-09-30 (Actual)

PRIMARY OUTCOMES:
PCR rate | 1 year
  pathological complete remission rate in T4NxM0 colorectal cancer treated after mFOLFOX6+Bevacizumab+PD-1monoclonal antibody

SECONDARY OUTCOMES:
Incidence rate of Grade ≥3 PD-1monoclonal antibody-related adverse events | 1 year
  Incidence rate of participants with Grade ≥3 PD-1monoclonal antibody-related adverse events as assessed by CTCAE v4.0
Incidence rate of Grade ≥3 chemotherapy-related adverse events | 1 year
  Incidence rate of participants with Grade ≥3 chemotherapy-related adverse events as assessed by CTCAE v4.0
R0 resection rate | 1 year
  R0 resection rate in participants treated after mFOLFOX6+Bevacizumab+PD-1monoclonal antibody
Down-stage rate | 1 year
  Down-stage rate of pathological stage after surgery compared with clinical stage before drug treatment
3 years DFS Rate | 3 years
  3 years Disease Free Survival Rate
3 years OS Rate | 3 years
  3 years Overall Survival Rate

CONTACTS AND LOCATIONS:
Overall Officials: Jun Huang, MD, Principal Investigator — Sixth Affiliated Hospital, Sun Yat-sen University
Locations (1):
- Sun Yatsen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Scott E. Chemohormonal therapy in metastatic hormone-sensitive prostate cancer. Sweeney CJ, Chen YH, Carducci M, Liu G, Jarrard DF, Eisenberger M, Wong YN, Hahn N, Kohli M, Cooney MM, Dreicer R, Vogelzang NJ, Picus J, Shevrin D, Hussain M, Garcia JA, DiPaola RS. Department of Medicine; Department of Biostatistics and Computational Biology; Dana-Farber Cancer Institute, Boston; Harvard Medical School, Boston; Johns Hopkins University, Baltimore; University of Wisconsin Carbone Cancer Center; School of Medicine and Public Health; Madison; Fox Chase Cancer Center, Temple University Health System, Philadelphia; Indiana University Melvin and Bren Simon Cancer Center, Indianapolis; Mayo Clinic, Rochester, MN; University Hospitals Case Medical Center, Seidman Cancer Center; Cleveland Clinic Taussig Cancer Institute; Both in Cleveland; University of Virginia Cancer Center, Charlottesville; Comprehensive Cancer Centers of Nevada, Las Vegas; Siteman Cancer Center, Washington University School of Medicine, St. Louis; NorthShore University Health System, Evanston, IL; University of Michigan Comprehensive Cancer Center, Ann Arbor; Rutgers Cancer Institute of New Jersey, New Brunswick.N Engl J Med. 2015 Aug 20;373(8):737-46. [Epub 2015 Aug 5]. doi: 10.1056/NEJMoa1503747. Urol Oncol. 2017 Mar;35(3):123. doi: 10.1016/j.urolonc.2016.12.021. Epub 2017 Feb 1. PMID 28159490
- [Result] Das R, Verma R, Sznol M, Boddupalli CS, Gettinger SN, Kluger H, Callahan M, Wolchok JD, Halaban R, Dhodapkar MV, Dhodapkar KM. Combination therapy with anti-CTLA-4 and anti-PD-1 leads to distinct immunologic changes in vivo. J Immunol. 2015 Feb 1;194(3):950-9. doi: 10.4049/jimmunol.1401686. Epub 2014 Dec 24. PMID 25539810
- [Result] Sclafani F. PD-1 inhibition in metastatic dMMR/MSI-H colorectal cancer. Lancet Oncol. 2017 Sep;18(9):1141-1142. doi: 10.1016/S1470-2045(17)30512-0. Epub 2017 Jul 19. No abstract available. PMID 28734760
- [Result] Antoniotti C, Borelli B, Rossini D, Pietrantonio F, Morano F, Salvatore L, Lonardi S, Marmorino F, Tamberi S, Corallo S, Tortora G, Bergamo F, Brunella DS, Boccaccino A, Grassi E, Racca P, Tamburini E, Aprile G, Moretto R, Boni L, Falcone A, Cremolini C. AtezoTRIBE: a randomised phase II study of FOLFOXIRI plus bevacizumab alone or in combination with atezolizumab as initial therapy for patients with unresectable metastatic colorectal cancer. BMC Cancer. 2020 Jul 22;20(1):683. doi: 10.1186/s12885-020-07169-6. PMID 32698790
- [Result] Bolhuis K, Kos M, van Oijen MGH, Swijnenburg RJ, Punt CJA. Conversion strategies with chemotherapy plus targeted agents for colorectal cancer liver-only metastases: A systematic review. Eur J Cancer. 2020 Dec;141:225-238. doi: 10.1016/j.ejca.2020.09.037. Epub 2020 Nov 12. PMID 33189037
- [Result] Chang H, Yu X, Xiao WW, Wang QX, Zhou WH, Zeng ZF, Ding PR, Li LR, Gao YH. Neoadjuvant chemoradiotherapy followed by surgery in patients with unresectable locally advanced colon cancer: a prospective observational study. Onco Targets Ther. 2018 Jan 17;11:409-418. doi: 10.2147/OTT.S150367. eCollection 2018. PMID 29398921
- [Result] Kim SA, Kim JW, Suh KJ, Chang W, Kim JW, Oh HK, Cho JY, Kim DW, Cho S, Kim JH, Kim K, Kang SB, Jheon S, Lee KW. Conversion surgery after cetuximab or bevacizumab plus FOLFIRI chemotherapy in colorectal cancer patients with liver- and/or lung-limited metastases. J Cancer Res Clin Oncol. 2020 Sep;146(9):2399-2410. doi: 10.1007/s00432-020-03233-7. Epub 2020 May 1. PMID 32358699
- [Result] Li J, Cong L, Liu J, Peng L, Wang J, Feng A, Yue J, Li L, Wang X, Wang X. The Efficacy and Safety of Regorafenib in Combination With Anti-PD-1 Antibody in Refractory Microsatellite Stable Metastatic Colorectal Cancer: A Retrospective Study. Front Oncol. 2020 Nov 12;10:594125. doi: 10.3389/fonc.2020.594125. eCollection 2020. PMID 33282742
- [Result] Marmorino F, Boccaccino A, Germani MM, Falcone A, Cremolini C. Immune Checkpoint Inhibitors in pMMR Metastatic Colorectal Cancer: A Tough Challenge. Cancers (Basel). 2020 Aug 17;12(8):2317. doi: 10.3390/cancers12082317. PMID 32824490
- [Result] Mise Y, Hasegawa K, Saiura A, Oba M, Yamamoto J, Nomura Y, Takayama T, Hashiguchi Y, Shibasaki M, Sakamoto H, Yamagata S, Aoyanagi N, Kaneko H, Koyama H, Miyagawa S, Shinozaki E, Yoshida S, Nozawa H, Kokudo N. A Multicenter Phase 2 Trial to Evaluate the Efficacy of mFOLFOX6 + Cetuximab as Induction Chemotherapy to Achieve R0 Surgical Resection for Advanced Colorectal Liver Metastases (NEXTO Trial). Ann Surg Oncol. 2020 Oct;27(11):4188-4195. doi: 10.1245/s10434-020-08627-y. Epub 2020 Jun 8. PMID 32514802
- [Result] Qiu B, Ding PR, Cai L, Xiao WW, Zeng ZF, Chen G, Lu ZH, Li LR, Wu XJ, Mirimanoff RO, Pan ZZ, Xu RH, Gao YH. Outcomes of preoperative chemoradiotherapy followed by surgery in patients with unresectable locally advanced sigmoid colon cancer. Chin J Cancer. 2016 Jul 7;35(1):65. doi: 10.1186/s40880-016-0126-y. PMID 27389519
- [Result] Yuan Y, Xiao WW, Xie WH, Cai PQ, Wang QX, Chang H, Chen BQ, Zhou WH, Zeng ZF, Wu XJ, Liu Q, Li LR, Zhang R, Gao YH. Neoadjuvant chemoradiotherapy for patients with unresectable radically locally advanced colon cancer: a potential improvement to overall survival and decrease to multivisceral resection. BMC Cancer. 2021 Feb 19;21(1):179. doi: 10.1186/s12885-021-07894-6. PMID 33607964